CLINICAL TRIAL: NCT00341185
Title: Studies of Thyroid Abnormalities in Northeastern Kazakhstan Associated With Nuclear Weapons Testing
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998014; OH98-C-N014
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-11-18

CONDITIONS: Thyroid Cancer
Keywords: Biodosimetry; Dose Reconstruction; Radioactive Fallout; Thyroid Screening; Ultrasound
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
We propose to study the prevalence of thyroid nodules and cancer in relation to radiation dose, in a defined cohort of Kazakhstan residents exposed as children to radioactive fallout from atomic bomb tests at the neighboring Semipalatinsk Test Site (STS). The population near the STS is believed to have received radiation doses from fallout that were much higher than that experienced by any population of comparable size in the US. The study population is a defined cohort of 20,000 residents, half of whom, in 1960, resided in heavily-exposed villages; the other half lived in lightly-exposed villages. The population is rural, with a diet that was and is heavily dependent upon fresh milk from household or local cows and therefore likely to have led to ingestion of radioactive iodine from fallout. The study is two parts.

The first part involves a cytogenetic assay for radiation biodosimetry purposes of peripheral lymphocytes obtained from blood samples donated by 40 cohort members with individuals radiation dose estimates. Blood samples will be collected from 25 putative high-dose and 15 low-dose cohort members and processed or cytogenetic assay using fluorescent in situ hybridization (FISH) for stable chromosome aberrations in peripheral lymphocytes. This biodosimetric validation assay, will be carried out by Nailya Chaizhunusova, chief of cytogenetics at the Scientific research Institute for Radiation Medicine and Ecology, in collaboration with Dr. Tracy Yang at the NASA Johnson Space Center in Houston, Texas. It should be possible to detect gamma radiation doses as low as 150 mGy.

The second part will involve thyroid screening by ultrasound in selected villages. The population to be screened will comprise 100-1500 members of the study cohort exposed as young children to high fallout levels, and equal numbers of comparable ages exposed to little or no fallout. Fine needle aspiration biopsy will be performed, under separate informed consent, if the palpation and ultrasound results suggest presence of a tumor. Presence and malignancy of tumor will be determined by cytopathology. Subjects with evidence of thyroid disease will be referred to thyroid specialists at the Semipalatinsk State Medical Academy. Finger stick blood samples will be obtained to assess thyroid function using RIA methods with coated tube technology for T4 and TSH. The most sensitive statistical comparisons are expected to be dose-response analyses with respect to prevalence of thyroid nodules, which are common and known to be associated with radiation dose. Comparisons in terms of thyroid cancer, and benign and malignant neoplasms combined, are likely to be less sensitive but of acceptable power if risks associated with chronic radiation in this population are similar to those associated with acute exposure to X-ray or gamma radiation in other populations.

DETAILED DESCRIPTION:
We propose to study the prevalence of thyroid nodules and cancer in relation to radiation dose, in a defined cohort of Kazakhstan residents exposed as children to radioactive fallout from atomic bomb tests at the neighboring Semipalatinsk Test Site (STS). The population near the STS is believed to have received radiation doses from fallout that were much higher than that experienced by any population of comparable size in the US. The study population is a defined cohort of 20,000 residents, half of whom, in 1960, resided in heavily-exposed villages; the other half lived in lightly-exposed villages. The population is rural, with a diet that was and is heavily dependent upon fresh milk from household or local cows and therefore likely to have led to ingestion of radioactive iodine from fallout. The study is two parts.

The first part involves a cytogenetic assay for radiation biodosimetry purposes of peripheral lymphocytes obtained from blood samples donated by 40 cohort members with individuals radiation dose estimates, and electron paramagnetic resonance (EPR) assays of about 110 stored tooth samples. The two techniques are complementary. Blood samples will be collected from 25 putative high-dose and 15 low-dose cohort members and processed or cytogenetic assay using fluorescent in situ hybridization (FISH) for stable chromosome aberrations in peripheral lymphocytes. This biodosimetric validation assay, will be carried out by Nailya Chaizhunusova, chief of cytogenetics at the Scientific research Institute for Radiation Medicine and Ecology, in collaboration with Dr. Tracy Yang at the NASA Johnson Space Center in Houston, Texas. It should be possible to detect gamma radiation doses as low as 150 mGy.

The EPR investigation will take advantage of a repository of teeth extracted by local dentists during medical and dental programs in 1966-67 and 1999, stored, and catalogued by our collaborators in Kazakhstan (not in connection with this study). Tooth samples are identified by village of exposure, but not individually within villages. However, the identities of the donors, and therefore their ages and exposure histories, are known to our collaborators in Kazakhstan; therefore it will be possible to compare the EPR results with gamma dose estimates calculated on the basis of exposure history. It is intended that the EPR assays will be carried out at the National Institute of Standards and Technology under a purchase order agreement.

The second part will involve thyroid screening by ultrasound in selected villages. The population to be screened will comprise 1000-1500 members of the study cohort exposed as young children to high fallout levels, and equal numbers of comparable ages exposed to little or no fallout. Fine needle aspiration biopsy will be performed, under separate informed consent, if the palpation and ultrasound results suggest presence of a tumor. Presence and malignancy of tumor will be determined by cytopathology. Subjects with evidence of thyroid disease will be referred to thyroid specialists at the Semipalatinsk State Medical Academy. Finger stick blood samples will be obtained to assess thyroid function using RIA methods with coated tube technology for T4 and TSH. The most sensitive statistical comparisons are expected to be dose-response analyses with respect to prevalence of thyroid nodules, which are common and known to be associated with radiation dose. Comparisons in terms of thyroid cancer, and benign and malignant neoplasms combined, are likely to be less sensitive but of acceptable power if risks associated with chronic radiation in this population are similar to those associated with acute exposure to X-ray or gamma radiation in other populations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be selected in accordance with the research aims of the project.

The majority should have whole-body or bone marrow radiation dose estimates as high as available among subjects who were children at the time of the major fallout events.

Few presumably low-exposure subjects are needed as null controls.

All subjects should have been born between 1940 and 1948.

EXCLUSION CRITERIA:

Subjects must not have a medical history including radiation therapy or high-dose diagnostic radiography or been treated for cancer.

Ages: 63 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2997 (Actual)
Dates: Start 1998-03-05; Study Completion 2016-11-18

PRIMARY OUTCOMES:
Thyroid Nodules | 1998

CONTACTS AND LOCATIONS:
Overall Officials: Kiyohiko Mabuchi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Semipalatinsk State Medical Academy, Semipalatinsk, Kazakhstan

REFERENCES:
- [Background] Hall P, Holm LE. Cancer in iodine-131 exposed patients. J Endocrinol Invest. 1995 Feb;18(2):147-9. doi: 10.1007/BF03349726. No abstract available. PMID 7629384
- [Background] Gusev BI, Abylkassimova ZN, Apsalikov KN. The Semipalatinsk nuclear test site: a first assessment of the radiological situation and the test-related radiation doses in the surrounding territories. Radiat Environ Biophys. 1997 Sep;36(3):201-4. doi: 10.1007/s004110050072. PMID 9402637
- [Background] Laird NM. Thyroid cancer risk from exposure to ionizing radiation: a case study in the comparative potency model. Risk Anal. 1987 Sep;7(3):299-309. doi: 10.1111/j.1539-6924.1987.tb00465.x. PMID 3685539